CLINICAL TRIAL: NCT06757660
Title: Effect of Two Irrigation Protocols Applied Prior to Furcation Repair on Post Operative Pain and Healing (A Randomized Clinical Trial)
Brief Title: Effect of Two Irrigation Protocols Applied Prior to Furcation Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shreef Mostafa Ibrahim, Assistant lecturer of Endodontics at Deraya University, minia, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shreef Mostafa
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2023-10

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 20 patients will be irrigated with Sodium hypochlorite (NaOCL 2.5%).using a negative pressure irrigation system to minimizes the risk of irrigant extrusion into the furcation space.
  Interventions: Procedure: Furcation Repair
- Group B (Active Comparator): About 20 patients will be irrigated with nanoparticle chitosan (2 %).
  Interventions: Procedure: Furcation Repair

INTERVENTIONS:
Procedure: Furcation Repair — to evaluate the clinical and radiographic effects of chitosan and Naocl as an irrigation protocols applied during repair of furcation perforation.

SUMMARY:
Perforations are mishaps that might occur during the course of endodontic treatment mainly due to iatrogenic factors. However, they might also occur due to extensive decay of dentinal structure.

A perforation creates a pathological passage between the root canal system and the periodontium and jeopardizes the success of the endodontic therapy. The damage caused by the perforation may eventually result in the extraction of the compromised tooth

DETAILED DESCRIPTION:
Chitosan is the most abundant biopolymer on the earth derived from chitin. It shows a remarkable effective broad spectrum antibacterial action attributed to its cationic nature. It interacts with the -ve charged bacterial cell membranes, leading to leakage of the intracellular constituents and ultimately cell death due to increasing the membrane permeability. Also, chitosan possesses a variety of other biological properties as being biodegradable, biocompatible and has chelating abilities, making it an interesting alternative to modern root canal irrigants.

Inadequacy of the repair materials has been a contributing factor to the poor outcome of repair procedures. On the basis of the recent physical and biologic property studies of the relatively new introduced mineral trioxide aggregate, this material may be suitable for closing the communication between the pulp chamber and the underlying periodontal tissues. There are few reports on repair of furcal perforation with MTA in molar teeth.

Several studies have stated the ability of chitosan as a chelating agent that potentially enhance the dentin wettability. At the same time, chitosan nanoparticles showed the potential to stabilize dentine collagen by providing resistance to bacterial collagenase degradation.

The null hypothesis: there is no difference in pain and healing between the two irrigation protocols of old fural perforations prior to application of Bio C repair material.

ELIGIBILITY:
Inclusion Criteria:

* Patients with old furcation perforation of mandibular molar.
* Size of perforation should be of average 1 to 2 mm.
* Period till treatment should be done within one month.
* Presence of polyp at the site of perforation is required in this study.

Exclusion Criteria:

* Teeth in need for post retained restoration.
* Immunocompromised patients.
* Pregnant women and smokers.
* Patients with a history of antibiotic or analgesics intake within the few days before the intervention and cases with previously initiated endodontic treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | From 1 day to 7 days after The Procedure
  Post-operative pain will be measured by a numerical pain rating scale (NRS), where the level of pain will be recorded as follows: 0 reading represents "no pain" ; 1- 3 reading represents "mild pain" ; 4- 6 reading represents "moderate pain" and 7- 10 reading represents "severe pain".

SECONDARY OUTCOMES:
Healing | From base line to 3,6 and 9 months
  Furcation repair development will be evaluated by comparing the furcation radiolucency, pre-operatively and postoperatively (after3, 6 and 9 months), using periapical radiographs and CBCT. This will be aggregated in percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Ali Moukarab, Professor, Study Chair — Endodontics,Faculty of Dentistry, Minia University; Esam Fawzy, Lecturer, Study Director — Department of Endodontics, Faculty of Dentistry Minia University
Locations (1):
- Minia University, Faculty of Dentistry, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided